CLINICAL TRIAL: NCT03399422
Title: Evaluation the Efficacy of Injectable Platelet Rich Fibrin (i-PRF) in Upper Canine Retraction and the Levels of Acceptance and Discomfort
Brief Title: Efficacy of Biological Technique in Upper Canine Retraction and Levels of Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-02-2018
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Malocclusion, Angle Class II, Division 1
Keywords: i-PRF (injectable platelet rich fibrin); canine retraction; pain and discomfort
MeSH Terms: conditions — Malocclusion, Angle Class II; Pain

STUDY DESIGN:
Intervention Model Description: Two Arms injectable platelet rich fibrin group: consisted of two subgroups
  Experimental group : injectable platelet rich fibrin assisted upper canine retraction Control group: conventional upper canine retraction
Who Masked: Outcomes Assessor
Masking Description: One blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF assisted upper canine retraction (Experimental): I-PRF assisted upper canine retraction will be performed in one side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars
  Interventions: Biological: i-PRF; Procedure: canine retraction
- conventional upper canine retraction (Experimental): Conventional upper canine retraction will be performed in the other side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars
  Interventions: Procedure: canine retraction

INTERVENTIONS:
Biological: i-PRF — i-PRF (injectable platelet rich fibrin) assisted upper canine retraction
  Arms: i-PRF assisted upper canine retraction
Procedure: canine retraction — upper canine retraction will be performed in one side of patients with Class II Division 1 malocclusion patients requiring therapeutic extraction of the maxillary first premolars

SUMMARY:
Twenty patients need therapeutic extraction of the maxillary first premolars with subsequent retraction of the maxillary canines, will be divided randomly into two groups, and will randomly assigned to one side of the maxillary arch at the first premolar region , and the other side served as the control. canine retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side , soldered transpalatal arch will be used as an anchor unit.

Pre- and post distalization dental casts will be evaluated to study rate of canine distalization, over a follow-up period until a Class I canine relationship will be achieved. The levels of Pain and discomfort will be monitored using a questionnaire with a VAS scale administered three times during the first day after prf injection.

DETAILED DESCRIPTION:
Reduced orthodontic treatment duration is important for care providers and orthodontic patients.it is also desirable that aesthetic concerns and time dependent adverse events such as discomfort, pain, external root resorption, suboptimal oral hygiene, white spot lesions and dental caries are held to the minimum. Although the surgical assisted accelerated orthodontic tooth movement (such as distraction of periodontal ligament, distraction of dentoalveolus, periodontally accelerated osteogenic orthodontics (PAOO),Corticision, orthognathic surgery, piezocision, piezopuncture and micro osteoperforation). It has been proved to be the most effective one currently, its disadvantages are: it is a bone surgery, and it causes loss of alveolar bone that undermines the periodontal support of the target teeth.

Noninvasive and nonsurgical methods have always been preferred by both the clinicians and the patients. These techniques have ranged from application of biological molecules to innovative technologies such as resonance vibration, cyclic forces, light electrical currents, magnetic field forces, low-intensity laser irradiation and low-level light therapy. Endogenously produced biologicals have been tested based on their roles in the turnover of alveolar bone in response to orthodontic tooth movement as well as during wound healing.

That's why the submucosal injection of platelet rich plasma (PRP) is a technique developed for accelerating orthodontic tooth movement by simulating the effects of bone insult without surgery and loss of alveolar bone, Some researchers found that prp injection created a regional acceleratory phenomenon-like effect which forms the basis of rapid tooth movement compared with conventional orthodontic treatment.

From here it has been thought about using a method to eliminate the surgical techniques' side effects. It has been found that platelet rich fibrin (PRF) has the ability to enhance tissue regeneration, accelerate wound healing and inducing stem cells differentiation through its growth factors (GFs).

PRF characteristics in comparison to platelet rich plasma PRP are:

1. its preparation is completely natural and there is no need for thrombin addition so there isn't immune reaction
2. it contains stem cells
3. it requires one stage centrifugation
4. PRF has been reported to gradually release autologous growth factors and expressed stronger and more durable effect on the cellular proliferation and differentiation than PRP in vitro This is the first study in the world that will use i-PRF with Orthodontic treatment, because of its benefits and easiness of using in dental clinic Study sample that consists of 20 patients, was calculated using (G-power sample size calculator), depending on the rate of canine retraction with a study power of 95%.

Allocation of the sides of intervention (PRF injection) and control sides is made by computer program (Excel).

After ensuring of the patients compliance with the terms and conditions of this study, the purpose and methods of the study will be explained to the patients using Information Sheet. In case of approval to participate, the patients asked to sign the Informed Consent.

Extra & Intra-oral photographs, impressions and clinical examination will be made.

Canine retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 150 g of force per side at the same time 20ml of patients' blood will be withdrawn and centrifuged (700 rpm within 3 minutes) to get 4ml i-PRF. PRF will be injected at the area of the extracted first premolar, The first point place is in the buccal interventional side (supra periosteal injection) and the second point place is in the palatal interventional side(sub periosteal injection). PRF will be injected twice at the beginning and at the middle of the canine retraction.

All measures will be analyzed before and after canine retraction between two sides.

A questionnaire will be given to the patients to study pain level accompanying PRF injection compared to the control side. Pain will be assessed using Visual Analogue Scale (VAS) 1 (No Pain) - 10 (Worst Pain).

A questionnaire will be given to the patients to study their acceptance of new treatment approach with comprehensive orthodontic treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 15-27 years.
2. Class II Division 1 malocclusion:

   Mild / moderate skeletal Class II (ANB ≤7) Overjet ≤10 Normal or excessive facial height (Clinically and then cephalometry assessed using these angles : SN-MP , MM , Y axis) Mild to moderate crowding ≤ 4
3. permanent occlusion.
4. Exist all the upper teeth (except third molars).
5. Good oral and periodontal health:

Probing depth < 4 mm No radiographic evidence of bone loss. Gingival index ≤ 1 Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, NSAIDs, …)
2. patients have anti indication for oral surgery ( medical - social - psycho)
3. Presence of primary teeth in the maxillary arch
4. Missing permanent maxillary teeth (except third molars).
5. Poor oral hygiene or Current periodontal disease:

   Probing depth ≥ 4 mm radiographic evidence of bone loss Gingival index > 1 Plaque index > 1
6. Patient had previous orthodontic treatment
7. Craniofacial anomalies (cleft lip and palate patients)
8. Smokers
9. coagulation disorders and patients treated with anticoagulants.
10. patients with immunodeficiency disorders

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change of the rate of canine retraction | Before the beginning of canine retraction and every 28 days until the canines will be in the proper position (class 1) which will be approximately after 6 months from the beginning of canine retraction
  The rate of canine retraction defines as the distance traveled in millimeters (mm) divided by the time required (in week).
  Orthodontic models will be taken before the beginning of canine retraction and every 28 days until the canines will be in the proper position (class 1).
  The distance of canine retraction will be calculated by measuring the difference between the initial cast and the final cast using the method described by Ziegler and Ingervall, which rely on Stable palatal reference Points (the medial ends of the third palatal rugae, Midpalatal Suture) and the tips of the canines and then this distance will be divided by the number of intervals (weeks) to give the rate of retraction in millimeters per week.
  Measurements will be made from the orthodontic models manually by direct technique using digital dental calipers.

SECONDARY OUTCOMES:
pain levels | on the first day after an hour, 2 hours and 6 hours of PRF injection
  A questionnaire will be given to the patients to study pain level accompanying PRF injection compared to the control side.
  Pain will be assessed using Visual Analogue Scale (VAS) 1 (No Pain) - 10 (Worst Pain)

CONTACTS AND LOCATIONS:
Overall Officials: Rania Haddad, PhD., Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Rosvall MD, Fields HW, Ziuchkovski J, Rosenstiel SF, Johnston WM. Attractiveness, acceptability, and value of orthodontic appliances. Am J Orthod Dentofacial Orthop. 2009 Mar;135(3):276.e1-12; discussion 276-7. doi: 10.1016/j.ajodo.2008.09.020. PMID 19268820
- [Background] Almpani K, Kantarci A. Nonsurgical Methods for the Acceleration of the Orthodontic Tooth Movement. Front Oral Biol. 2016;18:80-91. doi: 10.1159/000382048. Epub 2015 Nov 24. PMID 26599121
- [Background] Gulec A, Bakkalbasi BC, Cumbul A, Uslu U, Alev B, Yarat A. Effects of local platelet-rich plasma injection on the rate of orthodontic tooth movement in a rat model: A histomorphometric study. Am J Orthod Dentofacial Orthop. 2017 Jan;151(1):92-104. doi: 10.1016/j.ajodo.2016.05.016. PMID 28024792
- [Background] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Background] Naik B, Karunakar P, Jayadev M, Marshal VR. Role of Platelet rich fibrin in wound healing: A critical review. J Conserv Dent. 2013 Jul;16(4):284-93. doi: 10.4103/0972-0707.114344. PMID 23956527
- [Background] Ziegler P, Ingervall B. A clinical study of maxillary canine retraction with a retraction spring and with sliding mechanics. Am J Orthod Dentofacial Orthop. 1989 Feb;95(2):99-106. doi: 10.1016/0889-5406(89)90388-0. PMID 2916474
- [Derived] Zeitounlouian T, Haddad R, Brad B, Ballouk MA, Fudalej P. Does the application of autologous injectable Platelet-Rich Fibrin (i-PRF) affect the patient's daily performance during the retraction of upper canines? A single-centre randomized split-mouth controlled trial. BMC Oral Health. 2023 Nov 17;23(1):872. doi: 10.1186/s12903-023-03646-z. PMID 37978474